CLINICAL TRIAL: NCT05440032
Title: Electrochemical Test of Leukocyte Esterase as a Marker for Periprosthetic Joint Infection
Brief Title: LE as a Marker for Periprosthetic Joint Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center for Innovation and Research Organization (Network)
Responsible Party: Sponsor
Other Study IDs: LE001
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Prosthetic-joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Synovial fluid testing with semi-quantitative leukocyte esterase test strip: Using a drop of synovial fluid, sample will be analyzed via the point-of-care device to measure amount of leukocyte esterase in the sample
  Interventions: Diagnostic Test: Semi-quantitative electrochemical leukocyte esterse test strip
- Synovial fluid testing with Roche Chemstrip: Using a drop of synovial fluid, sample will be analyzed via a urine test-strip to measure amount of leukocyte esterase in the sample
  Interventions: Diagnostic Test: Roche Chemstrip

INTERVENTIONS:
Diagnostic Test: Semi-quantitative electrochemical leukocyte esterse test strip — Electrochemical assay to detect level of leukocyte esterase in sample
  Groups: Synovial fluid testing with semi-quantitative leukocyte esterase test strip
Diagnostic Test: Roche Chemstrip — Urinalysis chemstrip
  Groups: Synovial fluid testing with Roche Chemstrip

SUMMARY:
Testing and comparison of a novel point-of-care electrochemical assay to detect and help diagnose periprosthetic joint infection on the hip and knee to the standard of care test

DETAILED DESCRIPTION:
The primary objective of this study is to assess the equivalence of a semi-quantitative electrochemical leukocyte esterase test system and off-label use of the Roche Chemstrip leukocyte esterase (LE) test for the diagnosis of periprosthetic joint infection (PJI) in synovial fluid from hip and knee joints. In this study, the qualitative outcome of each of the two methodologies for detecting leukocyte esterase enzyme will be compared. The hypothesis of this study is that the two tests will demonstrate equivalence. The leukocyte esterase enzyme level will also be compared to synovial white blood cell count, which will be considered as a secondary reference.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Willing and able to sign the informed consent document
3. Subjects presenting with presumed aseptic failure of a prosthetic joint and expected to undergo revision arthroplasty, or subjects presenting with presumed PJI and expected to undergo either DAIR or radical implant resection, and subjects being investigated for PJI having joint aspiration outside of the operating room who may or may not require surgical intervention.

Exclusion Criteria:

1. Subjects with known active crystalline deposition disease (e.g. gout)
2. Subjects with adverse local tissue reaction (ALTR) as a result of corrosion of components or metal-on-metal bearing surface in the hip
3. Subjects with active inflammatory arthropathy (e.g. rheumatoid arthritis)
4. Subjects undergoing a second-stage re-implantation procedure for PJI
5. Subjects in which standard of care assessments, at a minimum serology (ESR and CRP) and synovial fluid analysis (synovial WBC count, neutrophil percentage, and culture), cannot be performed.
6. Subjects in whom there is an insufficient amount of synovial fluid to perform the required investigational tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing planned aseptic revision surgery to replace part or all of their hip or knee implant or subjects undergoing planned revision for infection
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Qualitative agreement (Positive, Intermediate, or Negative) between the semi-quantitative electrochemical LE test and Roche Chemstrip® LE test (Negative, Trace, 1+, or 2+) | Within one hour of fluid aspiration

SECONDARY OUTCOMES:
Correlation of leukocyte esterase and synovial white blood cell count | Within 30 days of surgery

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Colorado Joint Replacement, Denver, Colorado
  - Cleveland Clinic Florida, Weston, Florida
  - University of Louisville, Louisville, Kentucky
  - New York University, New York, New York
  - University of Rochester, Rochester, New York
  - JIS Orthopaedics, New Albany, Ohio
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - West Virginia University, Morgantown, West Virginia